CLINICAL TRIAL: NCT03767101
Title: Positive Affect and Mental Imagery in the Process of Cognitive Behavioural Therapy: the PACIfIC-Study
Brief Title: Positive Affect and Mental Imagery in the Process of Cognitive Behavioural Therapy
Acronym: PACIfIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ulrike Willutzki (Other)
Responsible Party: Sponsor-Investigator, Ulrike Willutzki, Clinical Professor, University of Witten/Herdecke
Organization: University of Witten/Herdecke (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 128/2018
Record Dates: First submitted 2018-11-26; First posted 2018-12-06 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Mental Disorders
Keywords: Positive affect; Mental imagery; Cognitive Behavioral Therapy; Psychotherapy process; Micro-intervention
MeSH Terms: conditions — Mental Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU + Positive mental imagery (Experimental): In all conditions the first eight sessions of treatment are focused. All sessions start with a brief, audio-tape presented positive mental imagery intervention (duration about six minutes). In this intervention patients are guided to imagine a happy, positive situation within the last seven days. Patients get the instruction to imagine from a field perspective, exploring various sensory modalities and feelings in that specific moment. Patients perform this task in the rooms of the treatment center together with their therapists. The text of the mental imagery intervention is standardized and spoken by Prof. Dr. Ulrike Willutzki. Directly before and after the imagination patients are asked on their mood with a single-item. After the short intervention patients are instructed to communicated the content of their imagination with their therapists for about one minute. After completion the regular cognitive behavioral therapy session begins.
  Interventions: Behavioral: Cognitive behavioral therapy
- TAU + Neutral mental imagery (Active Comparator): In all conditions the first eight sessions of treatment are focused. All sessions start with a brief, audio-tape presented neutral mental imagery intervention (duration about six minutes). In this intervention patients are guided to imagine a all-day, non-emotional provoking situation within the last seven days. Patients get the instruction to imagine from a field perspective, exploring various sensory modalities in that specific moment. Patients perform this task in the rooms of the treatment center together with their therapists. The text of the mental imagery intervention is standardized and spoken by Prof. Dr. Ulrike Willutzki. Directly before and after the imagination patients are asked on their mood with a single-item. After the short intervention patients are instructed to communicated the content of their imagination with their therapists for about one minute. After completion the regular cognitive behavioral therapy session begins.
  Interventions: Behavioral: Cognitive behavioral therapy
- Treatment as usual (Other): In all conditions the first eight sessions of treatment are focused. No additional intervention is conducted at the start of therapy sessions. Standard cognitive behavioral therapy is conducted during the whole treatment sessions.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — In all three treatment arms, licensed therapists/trainee therapists perform a cognitive behavior therapy (CBT) under conditions of the German health care system. All treatments are based on individualized treatment plans for each patient. Therapists are supervized by an CBT expert therapist in the outpatient treatment center. On average every forth session is supervized. The total duration of treatment is variable, oriented on patients symptoms and treatment goals.

SUMMARY:
Background: Research findings suggested that people with mental disorders show a dysfunctional upregulation of negative affect (NA) but at the same time a dysfunctional downregulation of positive affect (PA) as distinct processes. Nevertheless, established treatment approaches focus on the modification of problems and negative affect only. Experimental paradigms with healthy and subclinical populations showed that PA inductions lead to higher flexibility in information processing, cognitive appraisal and action tendencies. Higher amounts of PA were associated with more personal resources, higher psychological resilience and subjective well-being. Preliminary evidence indicated that a focus on positive and functional aspects in the life of patients lead to better treatment sessions and outcome. However, the role of PA for the process in cognitive behavioral therapy remains unclear.

Method/Design: In regard to this we developed the PACIfIC-study, serving the following objectives:

(1) to explore the trajectories of PA and NA and their association with relevant process variables in an early phase of CBT treatment. (2) To develop and test the feasibility of a brief and easily implementable intervention to promote PA in psychotherapy sessions. (3) To analyze the impact of this intervention on the therapeutic process between and within CBT sessions and intermediate outcomes.

The study includes a randomized contolled, longitudinal design in an outpatient research and treatment center. Both a process and an intervention analysis will be conducted. In the process analysis, we will examine the course of PA and NA in the first twelve sessions of CBT treatments. In the intervention analysis, we will examine the effects of a six-minute positive mental imagery intervention during an early phase of psychotherapy. The aim of this micro-intervention is to foster patients' in-session PA, which may lead to increased levels of subjective resources, resilience, and self-esteem (theory-driven outcome) as well as improvements in psychopathology and working alliance (secondary outcome).

Discussion: The study results may have important theoretical and practical implications on the use of PA in psychotherapeutic treatment. Furthermore an economic implementation of strengths-oriented interventions in psychotherapy practice may be initiated.

ELIGIBILITY:
Inclusion Criteria:

* at least one mental disorder according to DSM-5 criteria
* treatment at the center of Mental Health and Psychotherapy, Witten/Herdecke University; outpatients clinic

Exclusion Criteria:

* current diagnosis of a severe episode of major depressive disorder
* suffering from a psychotic disorder
* suffering from substance use disorder
* current episode of (hypo)mania
* current suicidal risk
* extensive experiences with guided mental imagery intervention
* insufficient German language skills
* currently receiving another psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) -session questionnaire- | Baseline; measured once per week for twelve weeks of treatment, directly after each session
  Outcome of the process analysis. International used self-report of positive and negative affect [20 items]. Participants will be asked to rate the items according to how they feel "in the current moment". Two subscales of global positive affect (ten items, range: 1-5) and global negative affect (10 items, range: 1-5) will be used separately. Subscale scores will be computed with averaged item scores.
Witten Resource Questionnaire (WIRF) -change measurement- | Baseline, mid-4 (after four weeks), mid-8 (after eight weeks), post-12 (after twelve weeks of treatment)
  Outcome of the intervention analysis. Self-report of psychosocial resources [subscale with 12 items]. A total score will be computed with averaged item scores (range: 0-5).
Connor-Davidson Resilience Scale (CD-Risc) -change measurement- | Baseline, mid-4 (after four weeks), mid-8 (after eight weeks), post-12 (after twelve weeks of treatment)
  Outcome of the intervention analysis. Internationally used self-report of psychological resilience [short version: 10 items]. A total score will be computed with averaged item scores (range: 1-7).
Rosenberg Self-esteem Scale (RSES) -change measurement- | Baseline, mid-4 (after four weeks), mid-8 (after eight weeks), post-12 (after twelve weeks of treatment)
  Outcome of the intervention analysis. Internationally used self-report of general self-esteem [10 items]. A total score will be computed with summed item scores (range: 0-30).

SECONDARY OUTCOMES:
Brief Symptom Inventory (BSI) -change measurement- | Baseline, mid-4 (after four weeks), mid-8 (after eight weeks), post-12 (after twelve weeks of treatment)
  Outcome of the intervention analysis. Internationally used self-report of symptom severity of patients [53 items].
Working Alliance Inventory - Short Revised (WAI-SR) -change measurement- | Baseline, mid-4 (after four weeks), mid-8 (after eight weeks), post-12 (after twelve weeks of treatment)
  Outcome of the intervention analysis. Internationally used self-report of therapeutic alliance measuring bond, goals and tasks in psychotherapy based on feedback of patients concerning the current therapy session [12 items].

OTHER OUTCOMES:
Resource-oriented Microprocess Analysis (ROMA) -Coding system of videotapes of treatment sessions with an observer rating- | In part video tapes of treatment sessions were analyzed; on average after two weeks, after five weeks and after eight weeks of treatment start
  Video-based coding system of different aspects of resource activation (resource units: personal resources, motivational resources, reframing of problems) and positive affectivity in treatment sessions on a minute-level in both patients and therapists. Videotapes are analyzed from an observer perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Willutzki, Prof. Dr., Study Chair — Witten/Herdecke University; Philipp Victor, Dr., Principal Investigator — Witten/Herdecke University
Locations (1):
- Witten/Herdecke University, Witten, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Schurmann-Vengels J, Fluckiger C, Reyer E, Odyniec P, Willutzki U. The Impact of Mental Imagery Instructions on Patients' and Therapists' Positive Affect and Strength-Based Behaviours Within Psychotherapy Sessions: A Randomized Controlled Process Study. Clin Psychol Psychother. 2024 Jul-Aug;31(4):e3036. doi: 10.1002/cpp.3036. PMID 39089326